CLINICAL TRIAL: NCT01488396
Title: Efficacy of 0.05% Cyclosporin Eye Drop in Stevens Johnson Syndrome Patient With Chronic Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pinnita Prabhasawat, Associated professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 336/2549
Record Dates: First submitted 2010-11-08; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Stevens-Johnson Syndrome
Keywords: Cyclosporin; Stevens-Johnson syndrome; Dry eye
MeSH Terms: conditions — Stevens-Johnson Syndrome; Dry Eye Syndromes | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.05%cyclosporin eye drop (Experimental)
  Interventions: Drug: 0.05%cyclosporin eye drop

INTERVENTIONS:
Drug: 0.05%cyclosporin eye drop — use twice daily for 6 months
  Other Names: cyclosporin A

SUMMARY:
The purpose of this study is to evaluate the efficacy of 0.05% cyclosporin ophthalmic emulsion (Restasis) in patients with Stevens-Johnson syndrome that have dry eyes by subjective symptoms and signs.

DETAILED DESCRIPTION:
Stevens-Johnson syndrome patients in chronic stage who have dry eys symptoms and signs will be treated with 0.05%cyclosporin ophthalmic emulsion(Restasis)twice a day for 6 months, compare results at 0,2,4,6 months include dry eye symptoms, corneal staining (Fluorescein, Rose Bengal), Schirmer I,FCT and impression cytology

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of legal age of consent
* Patient with Stevens-Johnson syndrome in chronic stage or has symptoms more than 3 months and has dry eye symptoms
* Dry eye symptoms are defined as

  1. has dry eye symptom everyday for more than 3 months
  2. has foreign body sensation frequently
  3. use tear substitutes more than 3 times per day
* Tear test shaw abnormalities at least 1 of 2 of following:

  1. Schirmer test without anesthesia is not more than 5 millimeters in 5 minutes
  2. Fluorescein clearance test at first 10 minutes is not more than 3 millimeters and has at least 1 of 3 of the following:

2.1.Rose Bengal score is not less than 4 2.2.Fluorescein stain at cornea 2.3.Impression cytology is consistent to dry eye

* Patent punctum

Exclusion Criteria:

* Age < 18 years old
* Patients with Steven Johnson syndrome without dry eye
* Patients used oral cyclosporine or anticholinergic drug within past 2 months
* Patients with HIV or immunocompromise status
* Patients with active ocular infections and patients with a history of herpes keratitis
* Patients with known or suspected hypersensitivity to any of the ingredients in the formula (cyclosporine, glycerin, castor oil, polysorbate 80, carbomer 1342)
* Female patients are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
dry eyes symptoms : dryness, gritty, photophobia, burning and pain | 0, 2, 4, 6 months

SECONDARY OUTCOMES:
Schirmer I test | 0, 6 months
Fluorescein clearance test (FCT) | 0, 6 month
Corneal staining | 0, 2, 4, 6 months
  Staining with fluorescein and rose bengal
Fluorescein tear break up time | 0, 2. 4. 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pinnita Prabhasawat, MD, Principal Investigator — Mahidol University
Locations (1):
- Mahidol university, Bangkok, Thailand